CLINICAL TRIAL: NCT02391987
Title: A Randomized Study of the Effectiveness of an Integrated Tele-monitoring and Patient-centric Health Coaching Strategy (Tele-HC) in Adult Patients Recently Hospitalized With Acute Decompensated Heart Failure (ADHF) Compared to Standard Care
Brief Title: Integrated Tele-monitoring and Patient-centric Health Coaching Strategy in Patients Hospitalized With Heart Failure
Acronym: Tele-HC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Preventice (Industry)
Responsible Party: Principal Investigator, Charles J. Bruce, Professor of Medicine, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-001448
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tele-Monitoring (Active Comparator): Tele-monitoring and health coaching in addition to standard health care
  Interventions: Device: Tele-monitoring and health coaching
- Standard Care (No Intervention): Standard care is defined as Heart Failure (HF) care based on current American College of Cardiology (ACC) and American Heart Association (AHA) HF guidelines implemented and orchestrated by a cardiologist and support staff at the participating institution.

INTERVENTIONS:
Device: Tele-monitoring and health coaching — Tele-monitoring involves a personal monitoring system used to analyze data to provide relevant health information back to the treating clinician and the user. The monitoring system remotely monitors electrocardiographic (ECG) signals, heart rate, breathing rate, and activity levels. Additional devices will be integrated with the monitoring device to assess blood pressure and weight.
  Health Coaching involves a team of health care professionals including a registered nurse (RN) . The health care team creates a plan specific to the patient and provides guidance on nutrition' medications, and exercise. The data collected by the remote monitoring device will assist the care team in patient management.
  Arms: Tele-Monitoring

SUMMARY:
This study evaluates the effectiveness of remote tele-monitoring and health coaching in helping to reduce hospitalizations in heart failure patients. Half of participants will receive tele-monitoring and health coaching, while the other half will receive standard health care provided by their chosen provider.

DETAILED DESCRIPTION:
Tele-monitoring involves a personal monitoring system used to analyze data to provide relevant health information back to the treating clinician and the user. The monitoring system remotely monitors electrocardiographic (ECG) signals, heart rate, breathing rate, and activity levels. Additional devices will be integrated with the monitoring device to assess blood pressure and weight.

Health Coaching involves a team of health care professionals including a registered nurse (RN). The health care team creates a plan specific to the patient and provides guidance on nutrition' medications, and exercise. The data collected by the remote monitoring device will assist the care team in patient management.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with primary or secondary diagnosis of Acute Decompensated Heart Failure (one or more of these symptoms: shortness of breath, orthopnea or edema AND one or more of these signs: rales, peripheral edema, ascites, or pulmonary vascular congestion on chest radiography)
* Adult patients >18 years old

Exclusion Criteria:

* Overall life expectancy < 1 year
* Known skin allergy to adhesives (hydrocolloid, silicone, acrylic)
* Active systemic infection
* Pregnant or lactating
* End stage renal disease on dialysis
* Subject or caregiver is not visually and tactile capable of smartphone and home device usage
* Inadequate cell phone coverage (including international patients or international travel during study period)
* Subject or legal guardian is not willing and able to provide appropriate informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-05; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bruce, MD, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Mayo Clinic, Jacksonville, Florida
  - Memorial Regional Medical Center, Mechanicsville, Virginia
  - St. Francis Medical Center, Midlothian, Virginia
  - St. Mary's Hospital, Richmond, Virginia
  - Mayo Clinic Health Systems, La Crosse, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Tele-Monitoring: Tele-monitoring and health coaching in addition to standard health care
  Tele-monitoring and health coaching: Tele-monitoring involves a personal monitoring system used to analyze data to provide relevant health information back to the treating clinician and the user. The monitoring system remotely monitors electrocardiographic (ECG) signals, heart rate, breathing rate, and activity levels. Additional devices will be integrated with the monitoring device to assess blood pressure and weight.
  Health Coaching involves a team of health care professionals including a registered nurse (RN) . The health care team creates a plan specific to the patient and provides guidance on nutrition' medications, and exercise. The data collected by the remote monitoring device will assist the care team in patient management.
Period: Overall Study
Arm/Group | Tele-Monitoring | Standard Care
Started | 54 | 58
Completed | 54 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tele-Monitoring | Standard Care | Total
Number analyzed (Participants) | 54 | 58 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (14) | 68 (13) | 69 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 63
  Male | 21 | 28 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 1 | 3
  Black or African American | 13 | 14 | 27
  White | 38 | 40 | 78
  Hispanic | 1 | 2 | 3
  Unknown or not reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 54 | 58 | 112

OUTCOME MEASURES:

1. Primary Outcome: Hospital Readmission
Description: Occurrence of all-cause hospital readmissions or death within 60 days
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-Monitoring | Standard Care
Number analyzed (Participants) | 54 | 58
Participants | 14 | 16
Statistical Analysis 1: Comparison: Tele-Monitoring vs Standard Care; Test type: Superiority; p = 0.73, Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of Readmissions or Visits
Description: Number of hospital readmissions or emergency room visits (visits without admissions)
Time Frame: 60 days
Measure: Number; unit: visits
Arm/Group | Tele-Monitoring | Standard Care
Number analyzed (Participants) | 54 | 58
visits | 19 | 20
Statistical Analysis 1: Comparison: Tele-Monitoring vs Standard Care; Test type: Superiority; p = 0.98, Cochran-Mantel-Haenszel

3. Secondary Outcome: Mortality
Description: All-cause mortality
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-Monitoring | Standard Care
Number analyzed (Participants) | 54 | 58
Participants | 1 | 4
Statistical Analysis 1: Comparison: Tele-Monitoring vs Standard Care; Test type: Superiority; p = 0.37, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to 60 days post discharge for all subjects
Arm/Group | Tele-Monitoring | Standard Care
All-Cause Mortality (participants affected / at risk) | 1/54 | 4/58
Serious Adverse Events (participants affected / at risk) | 2/54 | 2/58
Other Adverse Events (participants affected / at risk) | 5/54 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tele-Monitoring (N=54) | Standard Care (N=58)
Transient Ischemic Attack (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tiny Lacunar Infarct (Cerebral Vascular Accident) (Nervous system disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension and Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Shock Liver (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Right Heart Failure Exacerbation (Cardiac disorders) | 0 (0) | 1 (1)
Fluid overload (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tele-Monitoring (N=54) | Standard Care (N=58)
Wound at acrylic strip site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Reaction at acrylic strip site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Reaction at strip site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blisters in area having contact with strip (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blisters at acrylic/silicon strip site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT02391987/Prot_SAP_000.pdf